CLINICAL TRIAL: NCT02392390
Title: Effects of Topical Dynamic Phototherapy (TDP) on the Microbiota of Chronic Wounds: a Pilot Study
Brief Title: Effects of Topical Dynamic Phototherapy on the Microbiota of Chronic Wounds
Acronym: PDT-Bactério
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2014/LM-01; 2014-004668-40 (Other: RCB number)
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Leg Ulcer
Keywords: Topical Dynamic Phototherapy; Microbiota
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The study population (Experimental): A total of 10 leg ulcer patients will be recruted for this study. All will have the experimental treatment.
  Intervention: Topical Dynamic Phototherapy (TDP)
  Interventions: Procedure: Topical Dynamic Phototherapy (TDP); Drug: Metvixia cream

INTERVENTIONS:
Procedure: Topical Dynamic Phototherapy (TDP) — Metvixia cream is applied to the lesion (about 1mm thickness) and the treated zone is covered with an opaque dression for 3 hours. Any residual cream is removed an and the lesion immediately rinsed with saline solution when uncovering. One session (8 minutes) of phototherapy is then performed using an Altilite lamp in accordance with HAS (haute authorité de santé) recommendations.
Drug: Metvixia cream

SUMMARY:
The main objective of this study is to estimate the change in the relative numbers of commensal or low virulence potential bacteria before and after one session TDP.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

* To estimate changes in several microbiological parameters over three time periods (before treatment, after applying the Metvixia® and after irradiation during a single TDP session).
* Describe the evolution of the size and appearance of the wound 7d after the start of treatment
* Describe the potential adverse events associated with a TDP session

ELIGIBILITY:
Inclusion Criteria:

* Patient correctly informed concerning study implementation, objectives, constraints and patient rights
* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient presents with one or more leg ulcers (artieral, venous or mixed)
* Afebrile patient without periulcerous erythema and who does not require antibiotic therapy
* Patient who has not received antibiotic treatment during the last 7 Days

Nota bene: Patients with multiple ulcers at different stages will be included for the wound corresponding to the highest stage. If the patient has multiple ulcers atn the same stage, the deepest wound will be considered.

Exclusion Criteria:

* The patient is participating in another interventional study, has participated in another interventional study with the past 3 months, or is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has a contraindication for a treatment used in this study
* Patient with an infected leg ulcer treated with antibiotics
* Patients on curative anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The percentage of commensal or weak virulence potential bacteria among all bacteria species isolated per sample | Baseline (Day 0)
The percentage of commensal or weak virulence potential bacteria among all bacteria species isolated per sample | Day 0: immediately after Metvixia rinsing and right before phototherapy
The percentage of commensal or weak virulence potential bacteria among all bacteria species isolated per sample | Day 0: immediately after phototherapy

SECONDARY OUTCOMES:
The percentage of commensal bacteria among bacteria species isolated per sample | Baseline (Day 0)
The percentage of commensal bacteria among bacteria species isolated per sample | Day 0: immediately after Metvixia rinsing and right before phototherapy
The percentage of commensal bacteria among bacteria species isolated per sample | Day 0: immediately after phototherapy
The number of bacteria taxa detected per sample | Baseline (Day 0)
The number of bacteria taxa detected per sample | Day 0: immediately after Metvixia rinsing and right before phototherapy
The number of bacteria taxa detected per sample | Day 0: immediately after phototherapy
The diversity of bacteria taxa detected per sample (Shannon's H with log2) | Baseline (Day 0)
  Shannon's H with log2
The diversity of bacteria taxa detected per sample (Shannon's H with log2) | Day 0: immediately after Metvixia rinsing and right before phototherapy
  Shannon's H with log2
The diversity of bacteria taxa detected per sample (Shannon's H with log2) | Day 0: immediately after phototherapy
  Shannon's H with log2
The number of functional groups detected per sample | Baseline (Day 0)
  Function groups are predefined according to the presence/absence of each of the following factors: pathogen, anaerobic, cocci.
The number of functional groups detected per sample | Day 0: immediately after Metvixia rinsing and right before phototherapy
  Function groups are predefined according to the presence/absence of each of the following factors: pathogen, anaerobic, cocci.
The number of functional groups detected per sample | Day 0: immediately after phototherapy
  Function groups are predefined according to the presence/absence of each of the following factors: pathogen, anaerobic, cocci.
The diversity of functional groups detected per sample (Shannon's H with log2) | Baseline (Day 0)
  Shannon's H with log 2
The diversity of functional groups detected per sample (Shannon's H with log2) | Day 0: immediately after Metvixia rinsing and right before phototherapy
  Shannon's H with log 2
The diversity of functional groups detected per sample (Shannon's H with log2) | Day 0: immediately after phototherapy
  Shannon's H with log 2
Adverse events | Day 0
Adverse events | Day 7
Visual analog scale for pain during the phototherapy session | Day 0
  Scale from 0 to 10

OTHER OUTCOMES:
Age in years | Day 0 (baseline)
Gender | Day 0 (baseline)
Body mass index | Day 0 (baseline)
Number of lesions | Day 0 (baseline)
Initial wound care or follow up? | Day 0 (baseline)
If follow up visit, is the wound aggravated, stable or improving? | Day 0 (baseline)
If follow up visit, is the wound aggravated, stable or improving? | Day 7
Age of the target lesion in days | Day 0 (baseline)
Location of the target lesion | Day 0 (baseline)
  Heel, internal malleolus or external malleolus
Wound appearance | Day 0 (baseline)
  burgeoning, fibrinous, necrotic, blistering or de-epidermisation, exudative, bad odor
Presence/absence of signs of infection | Day 0 to Day 7
  Purulent discharge, local inflammatory signs, rough bony contact, associated osteitis without bone contact, bacteremia, severe sepsis
Change in the size of the wound (mm^2) | Day 7 versus baseline
Irradiation dose (minutes) | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Meunier, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France